CLINICAL TRIAL: NCT06992336
Title: A Phase II, Open-label, Randomized Trial to Compare Anlotinib and Immunotherapy and Capecitabine Versus Investigator's Choice Therapy in High Risk ctDNA Positive, Early Triple Negative Breast Patients With Residual Disease After Neoadjuvant Therapy
Brief Title: Circulating Tumor DNA Guided Boost Therapy in Early Triple Negative Breast Patients With Residual Disease After Neoadjuvant Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liu Qiang, Professor, Phd, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-281-01
Record Dates: First submitted 2025-04-29; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — anlotinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Experimental): Anlotinib 8mg qd PO，357days Benmelstobart 200mg i.v. Q3W or immunotherapy continued as in the NAC. Capecitabine 1000 或 1250 mg/m2 BID day1-14
  Interventions: Drug: Anlotinib ,; Drug: Benmelstobart; Drug: Capecitabine
- B (Active Comparator): Investigator's choice. If immunotherapy was used in the NAC setting, it was required to be used after NAC for up to 1 years.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Anlotinib , — Anlotinib 8mg qd PO，357days
  Arms: A
Drug: Benmelstobart — Benmelstobart 200mg i.v. Q3W
  Arms: A
Drug: Capecitabine — Capecitabine 1000 or 1250 mg/m2 BID day1-14

SUMMARY:
Early triple negative breast cancer patients who do not achieve pathologic complete response after neoadjuvant chemotherapy with or without immunotherapy have bad prognosis. ctDNA effectively identified patients with highest relapse risk.

This trial aims to explore whether the combination of anlotinib, immunotherapy and capecitabine could improve the outcome of this subgroup of high relapse risk patients compared with investigator's choice of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Stage II-III breast cancer patients, excluding occult breast cancer, inflammatory breast cancer, metaplasia breast cancer
* TNBC patients. TNBC was defined as ER <= 10%, PR <=10%, HER 0-1, or HER2 2+ and FISH negative.

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity is based on self-representation
Enrollment: 411 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2031-04-10 (Estimated); Study Completion 2036-01-01 (Estimated)

PRIMARY OUTCOMES:
iDFS | from randomization to any of the following events: local or distant relapse; contralateral breast caner, death of any cause，assessed up to 36 months.
  invasive disease free survival

SECONDARY OUTCOMES:
dDFS | from randomization to any of the following events: distant relapse; contralateral breast caner, death of any cause，assessed up to 36 months
  distant disease free survival
OS | from randomization to any of the following events: death of any cause，assessed up to 120 months
  overall survival
ctDNA clearance | From the time when post-operative ctDNA is tested to be positive to the time surveillence ctDNA turns negative, assessed up to 60 months
  the rate of patients whose ctDNA are positive after surgery and turns negative after boost therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangodng, China